CLINICAL TRIAL: NCT00095264
Title: A Study of Darbepoetin Alfa in Anemic Subjects With Low Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030207
Record Dates: First submitted 2004-11-02; First posted 2004-11-03 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa

SUMMARY:
The purpose of this study is to assess the effect of 13 weeks of darbepoetin alfa treatment on erythroid response in anemic subjects with low risk Myelodysplastic Syndrome (MDS).

ELIGIBILITY:
Eligibility Criteria: General: - Low risk MDS (low or intermediate-1 risk as defined by IPSS) and FAB classification of RA, RARS, or RAEB with blasts less than or equal to 10% determined via a bone marrow biopsy and CBC - Adequate iron stores determined by bone marrow film or section staining for iron via a bone marrow biopsy - ECOG Performance status score of 0, 1, or 2 Laboratory: - Local laboratory screening Hgb less than or equal to 11.0g/dL - Adequate renal function (serum creatinine concentration less than or equal to 2.0 mg/dL) - Adequate liver function (total bilirubin less than or equal to 2 times, ALT less than or equal to 3 times, and AST less than or equal to 3 times the upper limit of the respective normal range) Ethical: - Must be 18 years of age or older - Provide written Institutional Review Board (IRB)-approved informed consent before any screening procedures are performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209
Dates: Start 2004-10

PRIMARY OUTCOMES:
The proportion of subjects achieving an erythroid response during the 13-week test period

SECONDARY OUTCOMES:
The proportion of subjects achieving an erythroid response during the 28-week treatment period
The change in Hb from baseline
The incidence of red blood cell (RBC) transfusions (greater than or equal to 1 unit)
The change in FACT-F from baseline

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Gabrilove J, Paquette R, Lyons RM, Mushtaq C, Sekeres MA, Tomita D, Dreiling L. Phase 2, single-arm trial to evaluate the effectiveness of darbepoetin alfa for correcting anaemia in patients with myelodysplastic syndromes. Br J Haematol. 2008 Jul;142(3):379-93. doi: 10.1111/j.1365-2141.2008.07181.x. Epub 2008 Jun 6. PMID 18540943
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20030207.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/